CLINICAL TRIAL: NCT03678116
Title: Effects of Ingestion of a Commercially Available Thermogenic Dietary Supplement on REE, Cardiovascular, and Mood Responses
Brief Title: Effects of a Thermogenic Dietary Supplement on Metabolic, Hemodynamic, and Mood Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary Hardin-Baylor (Other)
Collaborators: Dymatize Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AMP-1
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Energy Metabolism; Heart Rate; Blood Pressure; Mood
Keywords: caffeine; metabolism
MeSH Terms: interventions — Sugars; Caffeine

STUDY DESIGN:
Intervention Model Description: Three groups: placebo, caffeine (plus Teacrine and Cayenne) and caffeine (plus Teacrine)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sugar Pill (Placebo) (Placebo Comparator): Taken with 8oz of water after baseline REE and hemodynamic measurements have been taken. One of three interventions to be consumed by the subjects. One week washout period required between treatments.
  Interventions: Drug: Sugar Pill (placebo)
- Caffeine (plus Teacrine and Cayenne) (Experimental): Taken with 8oz of water after baseline REE and hemodynamic measurements have been taken. One of three interventions to be consumed by the subjects. One week washout period required between treatments.
  Interventions: Dietary Supplement: Caffeine (plus Teacrine and Cayenne)
- Caffeine (plus Teacrine) (Experimental): Taken with 8oz of water after baseline REE and hemodynamic measurements have been taken. One of three interventions to be consumed by the subjects. One week washout period required between treatments.
  Interventions: Dietary Supplement: Caffeine (plus Teacrine)

INTERVENTIONS:
Drug: Sugar Pill (placebo) — Taken orally in capsule form
  Arms: Sugar Pill (Placebo)
Dietary Supplement: Caffeine (plus Teacrine and Cayenne) — Taken orally in capsule form
  Arms: Caffeine (plus Teacrine and Cayenne)
Dietary Supplement: Caffeine (plus Teacrine) — Taken orally in capsule form
  Arms: Caffeine (plus Teacrine)

SUMMARY:
This a randomized, double blind, placebo controlled, crossover design study which measures the effect of an available thermogenic dietary supplement on resting energy expenditure (REE), blood pressure and heart rate, and mood changes in moderate caffeine consumers. Participants will complete baseline measurements then ingest one of three pills. Once the pill is ingested, subjects will complete four REEs along with heart rate and blood pressure and appropriate questionnaires. Participants will return two more times, each after a one week washout period, and complete the same protocol with the remaining supplements.

DETAILED DESCRIPTION:
Subjects expressing interest in completing the study will be interviewed in the UMHB Human Performance Lab (HPL) to determine whether they qualify to participate in the study. Upon qualification, participants will be scheduled for their first testing session which will include: a body composition analysis via an InBody 770, hunger questionnaires, VAS questionnaires, follow up questionnaire, and 5 resting energy expenditure (REE) tests. Participants will be randomized into an order that determines which supplement to ingest at their testing sessions. Example: A, C, B will correspond to taking A the first session, C the second session and so on.

Supplementation protocol: Participants will be randomized into an order that determines which supplement to ingest at their testing sessions. Example: A, C, B will correspond to taking A the first session, C the second session and so on. Subjects will take one pill with 8oz of water in one minute of allotted time.

After initial REE, heart rate, blood pressure, questionnaires, and body composition tests, subjects will ingest the first of three supplements. After ingestion, subjects will complete four REEs every hour. At initial and 60 minutes post ingestion, ECG measurements will be recorded using the Biopac BSL. After each REE is complete, heart rate, blood pressure, and questionnaires will be taken and recorded. The REE will last 20 minutes, thus to ensure ending time is at the hour mark, the REE will be started at the 40 minute time point. Once testing is finished, subjects will return to the lab two more times with a one week washout period to ingest the remaining supplements.

Two days prior to each of the three testing sessions, participants will record their dietary intake via MyFitnessPal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be male or female between the ages of 18-35 years
* Subjects will not consume caffeine 24 hours prior to testing
* Subjects will be daily caffeine consumers (<200mg/day prior to 12pm)
* Subject has provided written and dated informed consent to participate in the study
* Subject is willing and able to comply with the protocol
* Subject is apparently healthy and free from disease, as determined by a health history questionnaire
* Subject agrees to log their diet 48 hours prior to each testing session
* Subject agrees to abstain from exercise 24 hours prior to each testing visit
* Subject agrees to fast for 12 hours prior to each testing visit
* Subject agrees to refrain from sleeping for one hour prior to and during each testing session

Exclusion Criteria:

* Subject has sensitivity issues following ingestion of caffeine
* Subject currently smokes or has quit within the last 6 months
* Subject takes medication prescribed by a physician or regularly takes over the counter medication
* Subject is allergic to any ingredient in the nutritional supplement or placebo
* Subject may be pregnant, is pregnant, is trying to become pregnant, or is breastfeeding
* Subject reports any unusual adverse events associated with this study that in consultation with the study investigators or their doctor recommends removal from the study
* Subject consumes >200 mg of caffeine before 12pm

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Effects of Ingestion of a Commercially Available Thermogenic Dietary Supplement on Resting Energy Expenditure (REE) | REE completed every hour for four hours post ingestion
  The primary purpose of this investigation is to determine the effectiveness of commercially available thermogenic dietary supplement on changing caloric expenditure via resting energy expenditure (REE) in daily, but modest caffeine consumers. This will be accomplished by observing caloric expenditure over a four hour time period post ingestion of the supplement as compared to baseline caloric expenditure pre-supplementation.
Effects of Ingestion of a Commercially Available Thermogenic Dietary Supplement on Heart Rate | Heart rate taken every hour for four hours post ingestion
  The primary purpose of this investigation is to determine the effectiveness of commercially available thermogenic dietary supplement on changing heart rate as measured by Omron HEM-907XL professional blood pressure monitor in daily, but modest caffeine consumers. This will be accomplished by observing heart rate over a four hour time period post ingestion of the supplement as compared to baseline heart rate pre-supplementation.
Effects of Ingestion of a Commercially Available Thermogenic Dietary Supplement on Blood Pressure | Blood pressure taken every hour for four hours post ingestion
  The primary purpose of this investigation is to determine the effectiveness of commercially available thermogenic dietary supplement on changes in both systolic and diastolic blood pressure as measured by Omron HEM-907XL professional blood pressure monitor in daily, but modest caffeine consumers. This will be accomplished by observing blood pressure over a four hour time period post ingestion of the supplement as compared to baseline blood pressure pre-supplementation.
Effects of Ingestion of a Commercially Available Thermogenic Dietary Supplement on Mood Responses | VAS values recorded every hour for four hours post ingestion
  The primary purpose of this investigation is to determine the effectiveness of commercially available thermogenic dietary supplement on changes in mood as measured by the Visual Analog Scale (VAS) in daily, but modest caffeine consumers. This will be accomplished by observing changes in mood over a four hour time period post ingestion of the supplement as compared to their baseline mood response pre-supplementation. The VAS measures levels of energy, focus, concentration, alertness, and fatigue.The VAS is used to measure attitudes over a continuum ranging from "lowest possible" to "highest possible". Participants are required to mark a line along a 10 centimeter line with one end titled "lowest possible" and the opposite end titled "highest possible". Scores for the scale range from 0 to 10 with levels of energy, focus, concentration, and alertness being towards the higher end of the scale, closer to 10. Levels of fatigue should be towards the lower end of the scale, closer to 0.

CONTACTS AND LOCATIONS:
Overall Officials: Lemuel W Taylor IV, PhD, Principal Investigator — UMHB Human Performance Lab
Locations (1):
- UMHB Human Performance Lab, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: No